CLINICAL TRIAL: NCT01752270
Title: The Effect of Diane-35 Pretreatment on Endocrine and Clinical Profile for Patients With Polycystic Ovary Syndrome Undergoing In-vitro Fertilization
Brief Title: the Effect of Diane-35 Pretreatment on In-vitro Fertilization Outcome for Patients With Polycystic Ovary Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Zhou Canquan, vice president, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sunyatsen8362
Record Dates: First submitted 2012-12-06; First posted 2012-12-19 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- diane-35 (Experimental): Diane-35 pretreatment from the third day of menstrual cycle
  Interventions: Drug: Diane-35 pretreatment
- blank control (No Intervention)

INTERVENTIONS:
Drug: Diane-35 pretreatment — Diane-35 is applied from the third day of menstrual cycle for 21 days with a 7-day interval, for 3 consecutive cycles.
  Arms: diane-35
Drug: Diane-35 pretreatment
  Arms: diane-35

SUMMARY:
Polycystic Ovary Syndrome is the most common endocrine disorder in women, is estimated to affect more than 5% of the population and is associated with chronically elevated serum androgen concentrations.Evidence suggests that polycystic ovary syndrome has a negative impact on pregnancy outcomes, with an increased risk of gestational diabetes, hypertensive disease during pregnancy,and preterm birth,which is partially related with the hyperandrogenic environment.Diane-35 has been proved to be the most effective anti-androgenic drug.At present, there is no direct evidence that Diane-35 has a positive effect on the clinical outcome of polycystic ovary syndrome patients undergoing In-vitro fertilization/Intracytoplasmic sperm injection.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed polycystic ovary syndrome patients according to Rotterdam criteria
* with hyperandrogenism and/or clinical hyperandrogenic manifestations
* no other oral contraceptives treatment for at least 3 months before this experiment
* no any other assisted reproductive therapy
* accompanied with fallopian tube and/or male factors
* normal hepato-/nephro- function

Exclusion Criteria:

* oral contraceptive pills contraindications, eg.Deep Venous Thrombosis
* smoking, drunk
* exclude other infertile factors, eg.endometriosis, abnormal thyroid function, etc.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
fertilization rate | up to 2years

SECONDARY OUTCOMES:
implantation rate | up to 2years

OTHER OUTCOMES:
clinical pregnancy rate | up to 2years

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun Yatsen University, Guangzhou, Guangdong, China